CLINICAL TRIAL: NCT04736810
Title: A Phase II Study of Penpulimab Combined With Chemotherapy ± Anlotinib Hydrochloride in Patients With Advanced Nasopharyngeal Carcinoma
Brief Title: A Study of Penpulimab Combination Therapy in Patients With Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akeso Tiancheng, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK105-205
Record Dates: First submitted 2021-01-30; First posted 2021-02-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Immunotherapy; Anti-PD-1 antibody; Nasopharyngeal Carcinoma; VEGF
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AK105 plus Gemcitabine and Anlotinib Hydrochloride (Experimental)
  Interventions: Biological: AK105; Drug: Cisplatin; Drug: Gemcitabine; Drug: Anlotinib hydrochloride

INTERVENTIONS:
Biological: AK105 — IV infusion
Drug: Cisplatin — IV infusion
Drug: Gemcitabine — IV infusion
Drug: Anlotinib hydrochloride — Oral administration

SUMMARY:
This is a multi-center, randomized, open-label, phase II study to evaluate the efficacy and safety of anti-PD-1 antibody Penpulimab (AK105) combined with chemotherapy ± anlotinib hydrochloride in the first-line treatment of patients with advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form voluntarily.
* Age over 18 years old (inclusive) and not more than 75 years old (inclusive), when signing the ICF.
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
* Expected life expectance ≥ 3 months.
* Histologically confirmed diagnosis of stage IVb NPC (AJCC 8th).
* Metastatic NPC patients who have not recieved the first-line platinumbased chemotherapy.
* At least one measurable tumor lesion per RECIST 1.1 criteria.
* Subjects must provide an available tumor tissue sample taken within 3 years prior to enrollment.
* Adequate organ function.
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception.
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use highly effective method of contraception from Day 1 and for 120 days after the last dose of investigational product.

Exclusion Criteria:

* Other invasive malignancies within 2 years, except for locally treatable (manifested as cured) malignancies, such as basal or skin squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ.
* Is currently participating in a study of an investigational agent or using an investigational device.
* Has known active central nervous system (CNS) metastases.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study.
* Has an active infection requiring systemic therapy.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment.
* Has undergone major surgery within 30 days of Study Day 1.
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 2 years
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) or death from any cause (whichever occurs first).
Disease control rate (DCR) | up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1.
Duration of response (DoR) | up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | up to 2 years
  OS is defined as the time from the date of randomization to death from any cause.
Observed concentrations of AK105 | From first dose of AK105 through 90 days after last dose of AK105.
  The endpoints for assessment of PK of AK105 include serum concentrations of AK105 at different timepoints after AK105 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK105 through 90 days after last dose of AK105.
  The immunogenicity of AK105 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Chen, MD, Study Chair — Cancer Hospital of The University of Chinese Academy of Sciences
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences, Hangzhou, Zhejiang, China